CLINICAL TRIAL: NCT01681758
Title: A Before-and-after Assessment of Pulse Pressure Variation Guided Fluid Therapy in Cardiac Surgery Patients Receiving Mandatory Mechanical Ventilation
Brief Title: An Assessment of Pulse Pressure Variation to Guide Fluid Therapy in Cardiac Surgery Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Austin Health (Other Government)
Responsible Party: Principal Investigator, Rinaldo Bellomo, Director of ICU Research, Austin Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AICU2012-007
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Cardiac Surgery
Keywords: cardiac surgery; Pulse pressure variation; intravenous fluids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PPV (Active Comparator): use PPV to guide fluid therapy
  Interventions: Other: IV fluid according to PPV
- standard care (Placebo Comparator): fluids according to standard care
  Interventions: Other: fluids according to standard care

INTERVENTIONS:
Other: IV fluid according to PPV — intravenous fluids
  Arms: PPV
Other: fluids according to standard care
  Arms: standard care

SUMMARY:
We aim to test the hypothesis that fluid therapy based on pulse pressure variation (PPV) in patients after cardiac surgery who are mechanically ventilated leads to a significant decrease in the amount of fluid given to such patients in the first 24 hours after surgery

DETAILED DESCRIPTION:
1. The investigators will study patients after cardiac surgery
2. The investigators will collect data on standard care in pre-intervention population
3. The investigators will collect demographic and clinical data
4. The investigators will collect biochemical data in the first 24 hours after surgery
5. The investigators will collect biochemical, physiological and clinical outcome data
6. The investigators will compare the standard care and intervention period data

ELIGIBILITY:
Inclusion Criteria:

1. immediately after ICU admission after cardiac surgery
2. mandatory mechanical ventilation -

Exclusion Criteria:

1. Pressure support ventilation
2. ECMO
3. Intra-aortic balloon counterpulsation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Mean amount of fluid given in the first 24 hours after surgery | 24 hours
  all intravenous fluid administered

SECONDARY OUTCOMES:
Physiological outcome | 24 hours
  Blood lactate

OTHER OUTCOMES:
Physiological outcome | 24 hours
  cardiac index

CONTACTS AND LOCATIONS:
Locations (1):
- Austin Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Suzuki S, Woinarski NC, Lipcsey M, Candal CL, Schneider AG, Glassford NJ, Eastwood GM, Bellomo R. Pulse pressure variation-guided fluid therapy after cardiac surgery: a pilot before-and-after trial. J Crit Care. 2014 Dec;29(6):992-6. doi: 10.1016/j.jcrc.2014.07.032. Epub 2014 Aug 7. PMID 25220528